CLINICAL TRIAL: NCT07126028
Title: Quality of Life in Children Who Were Treated for Multisystem Inflammatory Syndrome in Children
Brief Title: Quality of Life in Children After Multisystem Inflammatory Syndrome in Children
Acronym: MIS-C
Status: Enrolling by invitation | Type: Observational
Sponsor: Kristina Lah Tomulić (Other)
Responsible Party: Sponsor-Investigator, Kristina Lah Tomulić, assoc. prof., Clinical Hospital Center Rijeka
Organization: Clinical Hospital Center Rijeka (Other)
Other Study IDs: 003-05/22-1/93
Record Dates: First submitted 2025-08-02; First posted 2025-08-15 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Multisystem Inflammatory Syndrome in Children (MIS-C)
Keywords: risk adjustment; quality of life; Multisystem inflammatory Syndrome in Children
MeSH Terms: conditions — pediatric multisystem inflammatory disease, COVID-19 related

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MIS-C group: those children who survived MIS-C and were treated in the hospital
- control Group: healthy peers without any acute diseases or chronic conditions

SUMMARY:
The aim of this observational study is to assess whether Multisystem Inflammatory Syndrome (MIS-C) in children affects their quality of life. The investigators will examine whether there is a correlation between paediatric mortality prediction scoring systems, specific clinical and laboratory indicators, and whether some of these can predict the level of quality of life in children 24 months after hospital discharge.

The primary questions are:

Do children who survived MIS-C have a poorer quality of life 24 months after the illness compared to their peers? Can investigators identify prognostic indicators to create preventative strategies for MIS-C?

The investigator will compare the quality of life in participants who survived MIS-C with a control group. The quality of life will be measured using a validated questionnaire.

In the first phase, data from medical records will be collected. In the second, prospective part of the study, participants, healthy peers, and their parents or guardians will be asked to complete a questionnaire about quality of life.

DETAILED DESCRIPTION:
The COVID-19 pandemic has led to high morbidity and mortality in adults. Still, in children, the clinical picture and course of the disease are generally milder, and the overall estimated mortality rate is approximately 0.08%. However, it has been observed that in children after recovering from COVID-19, regardless of the severity of the clinical picture, a severe condition may occur, characterized by an inadequate hyper-inflammatory immune response with possible repercussions on various organ systems. Ultimately, the condition was recognised as a specific clinical entity which was named Multisystem Inflammatory Syndrome in Children (MIS-C). Guidelines for diagnosing a case of MIS-C have evolved. According to the current guidelines of the American Academy of Paediatrics, the following criteria must be met: 1. An individual aged <21 years and in the absence of a more likely alternative diagnosis; 2. Subjective or documented fever (T >38.0°C); 3. Clinical course requiring hospitalisation or leading to death; 4. C-reactive protein (CRP) >3.0 mg/dL; 5. New-onset manifestations that include >2 of the following categories: a) Cardiac: coronary artery dilation/aneurysm, left ventricular ejection fraction <55%, or troponin elevated above normal; b) Shock; c) Mucocutaneous: rash, oral mucosal inflammation, conjunctivitis/conjunctival injection, or extremity findings (erythema, edema); d) Gastrointestinal: abdominal pain, vomiting, or diarrhea; e) Hematologic: platelet count <150,000/µL, absolute lymphocyte count <1000/µL. 5. Detection of SARS-CoV-2 nucleic acid/antigen up to 60 days before or during hospitalisation or in a postmortem specimen, OR detection of antibodies associated with the current illness, OR close contact with a confirmed/probable case of COVID-19 within 60 days before hospitalisation. The clinical picture is very diverse, and most often affects the gastrointestinal, respiratory, cardiocirculatory, and haematological systems, as well as the skin and mucous membranes; however, any organ or organ system can be affected.

The therapeutic approach is based on the use of organ-specific supportive and immunomodulatory therapy. Treatment guidelines recommend the use of intravenous immunoglobulins (2 g/kg), then corticosteroids (2-30 mg/kg/day methylprednisolone, depending on the severity of the disease) and finally biological therapy (most often anakinra, 2-10 mg/kg/day), with thromboprophylaxis with aspirin. Although these are mostly previously healthy children, it is described in research that even up to 80% of them required treatment in JILD, and in certain patients, it led to death. Since in a large part of these patients there is involvement of the heart, which includes ventricular dysfunction, enlargement or aneurysm of the coronary artery and arrhythmias, there is a need for longer-term follow-up due to the unclear prognosis and the risk of progression of cardiac manifestations, and in a smaller number of patients, the persistence of cardiac dysfunction has been described even six months after discharge from the hospital. Although less common, neurological manifestations are part of the clinical picture of MIS-C and carry a significant risk of chronic morbidity and mortality; Neurological sequelae and long-term neurodevelopmental outcomes are currently unknown and require further research. Longer-term follow-up of children with MIS-C is of interest. Even in cases of recovery, given the broad spectrum of the disease, its involvement of nearly all organ systems, and the variable clinical presentation, there is a need for regular and continuous follow-up and contact with medical care.

Aim and Purpose of the Research This scientific research hypothesises that children suffering from MIS-C have a worse quality of life compared to their peers, as measured by validated HRQoL questionnaires, 24 months after hospital discharge.

The second hypothesis is that the value of the PRISM III/IV and PIM-3 scores in children suffering from MIS-C correlates with the outcome and quality of life measured 24 months after hospital discharge.

Specific research objectives:

1. To assess the quality of life of children treated for MIS-C 24 months after hospital discharge and correlate them with healthy peers of the same age and sex
2. To investigate the relationships between two scoring systems for predicting mortality and the quality of life of children 24 months after hospital discharge
3. To investigate whether any specific laboratory, clinical, or other indicators (such as length of hospitalisation, applied therapy, or comorbidity) can predict a poorer quality of life in children 24 months after hospital discharge.

Participants

In the first part of the study, the participants will be:

1. Children who have recovered from MIS-C All children suffering from and treated for MIS-C, who at the time of admission met the criteria for diagnosis, were admitted to the Pediatric Clinic of the Rijeka University Hospital Centre and the Clinic for Infectious Diseases "Dr. Fran Mihaljević", in the period from May 1, 2020, to April 30, 2022. The group planned for the study includes all children aged 1 month to 18 years treated in the institutions mentioned above, admitted during the period mentioned earlier, regardless of the severity of the clinical picture or possible comorbidities.

In the second part of the study, the participants will be:

1. All participants from the first group who survived MIS-C
2. A control group of healthy peers who will be compared with the first in such a way that each subject from the first group will be compared with one healthy subject of the same age and sex

Only children who do not meet any of the exclusion criteria and whose parents or legal guardians, or themselves (if older than twelve years of age), have signed an informed consent form will be included in the study. The exclusion criteria will be:

* all patients who died due to MIS-C
* refusal to participate in the study

Methods:

The first part of the study will include approximately 85 children. Data will be collected and stored in the hospital information system (BIS) within 24 hours of patient admission from recorded clinical and laboratory parameters that are part of routine processing when a patient is admitted to the ward. For each child in the specified period, the risk of mortality will be assessed using two different risk assessment scoring systems: PIM III (Pediatric Index of Mortality) and PRISM III/IV (Pediatric RISk of Mortality). The data will be entered into the existing program for calculating the mortality risk for each scoring system. The data will be entered at the Rijeka Clinical Hospital by the principal investigator and at the "Dr. Fran Mihaljević" Clinic by a pediatric infectious disease specialist, who is also a co-investigator in the research work. The data will be anonymous and entered into the database under a code.

In the second part of the study, the quality of life of all surviving children with MIS-C will be examined, for at least 24 months from discharge from the hospital, and compared with the quality of life of healthy children of the same age and sex to establish the credibility of the data obtained and enable the possibility of comparison. The quality of life will be examined using a questionnaire, which will be completed depending on age, by parents or guardians, and children over five years old. The questionnaire "Pediatric Quality of Life Inventory™ Generic Core Scales (PedsQL™ Generic Core Scales)" will be used. The questionnaire examines and obtains answers related to the areas of physical health and activity, emotional health, social activities and school/kindergarten activities. The answers obtained are reverse-scored and linearly transformed into a scale, so that higher scores indicate better quality of life. The questionnaire has been validated in both English and Croatian, and permission from the author has been obtained for its use in Croatian. Data will be collected by the principal investigator either during regular check-ups at the Clinic or by the responsible paediatricians. After regular check-ups for at least 24 months following discharge from MIS-C, all parents and children will be offered a questionnaire in the clinics, regardless of whether the child is chronically ill or healthy; that is, all children will be treated equally. The questionnaires are designed for a heterogeneous group of children and demonstrate exceptional reliability in distinguishing between healthy and acutely and chronically ill children. The control group will include healthy children of the same age and gender, without acute or chronic diseases. This means they have no history of acute hospitalisations in hospitals for any reason and no information on chronic health problems, including chronic childhood diseases and chronic physical disabilities. Examples of chronic diseases include, among others, childhood asthma, cystic fibrosis, congenital heart defects, diabetes, epilepsy, chronic inflammatory bowel disease, celiac disease, rheumatological diseases such as juvenile idiopathic arthritis, and psychiatric disorders (e.g., attention deficit hyperactivity disorder and depression).

The participants will be recruited by the primary care physician, who is also the responsible physician for the control patient treated by MISC, through random selection from the hospital records of children of the desired age. The responsible physician will then contact the parent of the potential healthy subject and offer them the opportunity to participate in the study. The time to complete the questionnaire is five to ten minutes. The obtained data will then be analysed to correlate the values of the mortality scoring system parameters with the quality of life assessment data and to determine whether a positive correlation can be observed.

ELIGIBILITY:
Inclusion Criteria:

* children of the same age and gender as the children in MIS-C group

Exclusion Criteria:

* history of acute hospitalisations in hospitals for any reason
* chronic health problems (including chronic childhood diseases and chronic physical disabilities)

Examples of chronic diseases include:

* childhood asthma
* cystic fibrosis
* congenital heart defects
* diabetes mellitus
* epilepsy
* chronic inflammatory bowel disease
* celiac disease
* rheumatological diseases such as juvenile idiopathic arthritis
* psychiatric disorders (e.g., attention deficit hyperactivity disorder and depression).

Examples of chronic physical disabilities include:

* hearing or vision impairment
* cerebral palsy
* myelomeningocele
* loss of limb function

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The subjects will be recruited by the primary care physician, who is also the responsible physician for the control patient treated by MIS-C, through random selection from the hospital records of children of the desired age. The responsible physician will then contact the parent of the potential healthy subject and offer them the opportunity to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To assess the quality of life of children with and treated for MIS-C 24 months after hospital discharge | from enrollment (24 weeks after hospital discharge) to the end of completing the questionnaire at 12 weeks
  The quality of life of all surviving children with MIS-C will be examined using a validated questionnaire for at least 24 months from discharge from the hospital.
  The quality of life will be assessed using a questionnaire completed based on age, by parents or guardians for children under five, and by children over five years old themselves. The questionnaire used is the "Pediatric Quality of Life Inventory™ Generic Core Scales (PedsQL™ Generic Core Scales)." It investigates and gathers responses related to physical health and activity, emotional health, social activities, and school or kindergarten activities.
  Each response can score between 0 and 4 points, where 0 indicates the best outcome and 4 the worst.
  The responses are reverse-scored and linearly transformed into a scale so that higher scores represent better quality of life (for 0 = 100, 1 = 75, 2 = 50, 3 = 25, and 4 = 0).
The quality of life of healthy peers | From enrollment to the end of completing the questionnaire at 12 weeks.
  A control group of peers (healthy participants) of the same age and sex will complete the questionnaire.
  The quality of life will be assessed using a questionnaire completed based on age, by parents or guardians for children under five, and by children over five years old themselves. The questionnaire used is the "Pediatric Quality of Life Inventory™ Generic Core Scales (PedsQL™ Generic Core Scales)." It investigates and gathers responses related to physical health and activity, emotional health, social activities, and school or kindergarten activities.
  Each response can score between 0 and 4 points, where 0 indicates the best outcome and 4 the worst.
  The responses are reverse-scored and linearly transformed into a scale so that higher scores represent better quality of life (for 0 = 100, 1 = 75, 2 = 50, 3 = 25, and 4 = 0).

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Hospital Centre Rijeka, Department of Paediatrics, Rijeka, Primorje-Gorski Kotar County, Croatia

IPD SHARING:
Plan to Share IPD: Yes
All information about the investigation plan: recruitment methods, statistics used in the study and results after completing the research.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: May 2026 - December 2026